CLINICAL TRIAL: NCT01986153
Title: Essential Fatty Acid Status & Immune Function in Parenteral Nutrition Patients
Status: Completed | Type: Observational
Sponsor: Geert Wanten (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Geert Wanten, MD, PhD, MSc, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Other Study IDs: 2013/475
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Intestinal Failure
Keywords: Fatty acid, essential; Immune system; Home parenteral nutrition
MeSH Terms: conditions — Intestinal Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Home parenteral nutrition patients: Patients who receive home parenteral nutrition.
- Healthy controls: Those who don't receive home parenteral nutrition and consume a normal diet.

SUMMARY:
The purpose of this study is to determine if patients on long-term olive oil-based parenteral nutrition have an adequate essential fatty acid status and immune status, compared to age- and sex-matched healthy controls.

DETAILED DESCRIPTION:
Patients, who suffer from severe chronic intestinal failure and whose nutritional intake cannot be met by oral food intake, have as their final option total parenteral nutrition, which contains all necessary macro- and micronutrients. Lipid emulsions are essential for these patients as they are a source of non glucose fuel calories, and they contain (essential) fatty acids which are important as structural component for many cells in the human body. Home parenteral nutrition patients are at risk for essential fatty acid deficiency. Data are lacking that indicate the optimal amount of essential fatty acids required for these patients. The latter seems especially relevant for patients receiving lipid prescriptions which are low in essential fatty acids, like ClinOleic®. Long-term parenteral nutrition dependent patients successfully use ClinOleic®. It is however unknown whether these patient remain to have an adequate essential fatty acid status in the long run.

ELIGIBILITY:
Home parenteral nutrition patients:

Inclusion Criteria:

* home parenteral nutrition: at least 6 months with a minimum frequency of 5 times a week

Exclusion Criteria:

* active immune modulating (underlying) disease
* use of immune suppressives
* use of oral fish oil substrates
* smoking more than 5 cigarettes/day
* do not eat more than 5 portions of fatty fish per week

Healthy controls:

Inclusion Criteria:

* age and sex matched healthy volunteer

Exclusion Criteria:

* active immune modulating (underlying) disease
* use of immune suppressives
* use of oral fish oil substrates
* smoking more than 5 cigarettes/day
* do not eat more than 5 portions of fatty fish per week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Long-term parenteral nutrition dependent patients:Patients who visit the outpatient clinic of the Department of Gastroenterology and Hepatology at the Radboud University Medical Nijmegen Center.
  Healthy controls: volunteers who are residents in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Essential fatty acid status of plasma phospholipids and peripheral blood mononuclear cells, including the biochemical determination of the Holman index (ratio of mead acid/ arachidonic acid) | On day of blood withdrawal

SECONDARY OUTCOMES:
Physical examination of clinical signs/symptoms of essential fatty acid deficiency | On day of blood withdrawal
Immune function: expression of cell surface markers, stimulus-induced reactive oxygen species production, cytokine production by leukocytes | On day of blood withdrawal

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology and Hepatology, Nijmegen, Netherlands